CLINICAL TRIAL: NCT01777477
Title: Gemcitabine Combined With Chloroquine in Patients With Metastatic or Unresectable Pancreatic Cancer. A Dose Finding Single Center Phase I Study
Brief Title: Adjuvant Effect of Chloroquine on Gemcitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONK-USZ-004
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chloroquine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chloroquin in addition to Gemcitabine (Experimental): Gemcitabine 1000 mg/m2 i.v. at days 1, 8, 15 of every 28-day cycle. Chloroquine 100 mg, 200 mg or 300 mg (according to dose level) p.o. at days 2, 9, 16 of every 28-day cycle.
  Interventions: Drug: Chloroquine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Chloroquine — Addition of Chloroquine to Gemcitabine
  Other Names: Nivaquin
Drug: Gemcitabine
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to evaluate the safety by defining the maximum tolerated dose (MTD) of Choloroquine when combined with Gemcitabine, and to evaluate preliminary efficacy of combined systemic Gemcitabine and Chloroquine. In addition, the influence of the treatment on the anti-cancer immunity and the value of GOLPH2 as serum marker for pancreatic cancer will be assessed within a translational objective.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed non-resectable locally advanced or metastatic adenocarcinoma of the pancreas. Assessment is done within 21 days before enrolment.
* Age = 18 years
* Adequate liver function or kidney function tests, including any of the following: Bilirubin < 2 x ULN, Alanin-Aminotransferase (ALT) < 5 x ULN, Alcaline phosphatase < 5 x ULN, Estimated creatinine clearance > 40 ml/min (using the Cockroft formula)
* Adequate haematological values: Haemoglobin > 80 g/L, Leukocytes >3.00 g/L, Neutrophils > 1.00 g/L, Platelets > 100 g/L
* Written informed consent
* Biliary decompression is mandatory before inclusion into the study in case of bilirubin levels > 50 µmol/L.
* Women who are not breastfeeding and are using effective contraception if sexually active, who are not pregnant and agree not to become pregnant during the 12 months thereafter. A negative pregnancy test before inclusion into the trial is required for women of childbearing potential, defined as having not reached the menopause, last menstrual period occurred less than 12 months ago, no surgical sterilization performed, and fallopian tubes and/or uterus have been not surgically removed.
* Men who agree not to father a child during participation in the trial or during the 12 months thereafter.

Patient compliance and geographic proximity allow proper staging and follow-up. Patient not eligible for FOLFIRINOX treatment. WHO PS 0-2

Exclusion criteria:

* Life expectancy < 3 months
* Severe medical or psychiatric co-morbidity prohibiting the planned treatment or the giving of informed consent
* Any prior chemotherapy for pancreatic cancer, including adjuvant chemotherapy.
* Any prior radiotherapy or combined radio-chemotherapy for pancreatic cancer if completed less than 12 months prior to study inclusion.
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
* Known glucose-6-phosphate dehydrogenase deficiency.
* Concurrent use of other experimental drugs, treatment within a clinical trial within 30 days prior to trial entry.
* Active heart disease defined as congestive heart failure > NYHA class 2
* Past or current history (within the last 2 years prior to treatment start) of other malignancies except basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Inability or unwillingness to comply with the study protocol
* No understanding of the german language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of orally administered Chloroquine with concomitant intravenous Gemcitabine. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Samaras, MD, Principal Investigator — University Hospital Zurich, Department of Oncology
Locations (1):
- University Hospital Zurich, Department of Oncology, Zurich, Canton of Zurich, Switzerland